CLINICAL TRIAL: NCT05235776
Title: New-onset Severe Headache After Covid-19 Vaccine
Acronym: CovaxHEAD
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other); Hodepineklinikken Bergen (Unknown); Molde Hospital (Other); Namsos Hospital (Other); Medi3 (Unknown); Oslo Hodepinesenter (Unknown); Sandvika Nevrosenter (Unknown)
Responsible Party: Principal Investigator, Anne Hege Aamodt, Dr., Oslo University Hospital
Other Study IDs: 351097
Record Dates: First submitted 2022-02-08; First posted 2022-02-11 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Headache; Migraine; COVID-19
MeSH Terms: conditions — Headache; Migraine Disorders; COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — observation

SUMMARY:
Hypotheses:

1. Severe new-onset headache after Covid-19 vaccine occur in a minor subset of vaccinated individuals.
2. Immunological reactivity with activation of trigeminal nociceptors can be among the mechanisms in severe headaches after Covid-19 vaccines.
3. Biomarkers in blood and CSF and imaging findings can be used to assess severe new-onset headache after Covid-19 vaccines.

The main aim of the project is to describe the characteristics of severe new-onset headache after Covid vaccine and the treatment effects.

Secondary aim:

1. Investigate potential mechanisms and analyse biomarkers to predict treatment effects.
2. To assess at baseline and 6-month follow-up the rate of brain MRI pathology.
3. To assess the change xof brain 18F-FDG PET metabolism from baseline and 6-month follow-up
4. To assess the levels of brain specific biomarkers
5. To assess the level of blood specific biomarkers

Duration of Study participation:

* Enrollment: 24 months
* Follow-up: at 3 and 6 months after inclusion. For those with continued severe headache regular 3-month controls are planned during the study.

Total study duration 24 months

DETAILED DESCRIPTION:
Study Design: Prospective observational multi-center study

Cohort study of patients with new-onset severe headache after Covid-19 vaccine. Patients referred to the participating headache clinics for severe headache after Covid vaccine will be invited to participate in the study. The invitation will be given in conjunction with their visit to the headache specialist. Patients already diagnosed and treated for severe headache after Covid vaccine will be invited to participate during control visits at the participating centres. After written informed consent information information from the initial phases will be collected retrospectively from the medical records of the patients that have already been diagnosed and started with treatment. Further information will be collected prospectively. For newly diagnosed patients all information will be collected prospectively. Blood samples will be drawn to assess immunological mechanisms.

Inclusion criteria:

* Patients aged ≥ 18 years with new onset severe headache or severe worsening of pre-existing headache within one week after Covid vaccination and has not resolved within 3 weeks.
* Inclusion within 12 months after symptom onset.
* Informed written consent signed by the patient.

Exclusion criteria:

• Patients not available for follow-up assessments (e.g. non-resident).

ELIGIBILITY:
IInclusion criteria:

* Patients aged ≥ 18 years with new onset severe headache or severe worsening of pre-existing headache within one week after Covid vaccination and has not resolved within 3 weeks.
* Inclusion within 12 months after symptom onset.
* Informed written consent signed by the patient.

Exclusion criteria:

• Patients not available for follow-up assessments (e.g. non-resident).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort study of patients with new-onset severe headache after Covid-19 vaccine. Patients referred to the participating headache clinics for severe headache after Covid vaccine will be invited to participate in the study. The invitation will be given in conjunction with their visit to the headache specialist. Patients already diagnosed and treated for severe headache after Covid vaccine will be invited to participate during control visits at the participating centres. After written informed consent information information from the initial phases will be collected retrospectively from the medical records of the patients that have already been diagnosed and started with treatment. Further information will be collected prospectively. For newly diagnosed patients all information will be collected prospectively. Blood samples will be drawn to assess immunological mechanisms
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Characteristics of the of new onset headache after Covid vaccination | at inclusion
  qualitative description
Characteristics of the of new onset headache after Covid vaccination | 6 months
  qualitative description

SECONDARY OUTCOMES:
Days with headache ((defined by headache intensity > 0 and/ patient's acute headache medication) | at inclusion
  number of days
Days with headache ((defined by headache intensity > 0 and/ patient's acute headache medication) | at 6 months
  number of days
Headache intensity (0-3 scale) on days with headache at baseline | at inclusion
  Headache intensity, number
Duration of new onset headache after Covid vaccination at baseline | at inclusion
  number of hours
Duration of new onset headache after Covid vaccination at 6 months follow-up | at 6 months
  number of hours
The six item Headache Impact Test (HIT-6) score at baseline | at inclusion
  HIT-6 score
The six item Headache Impact Test (HIT-6) score at 6 months follow-up | at 6 months
  HIT-6 score
The rate of brain MRI pathology at baseline | at inclusion
  description of MRI pathology
The change of brain 18F-FDG PET/CT metabolism | 6 months
  description of brain 18F-FDG PET/CT metabolism
The levels of brain specific biomarkers | at inclusion
  The levels of brain specific biomarkers
The level of blood specific biomarkers | at 6 months
  The levels of brain specific biomarkers

CONTACTS AND LOCATIONS:
Locations (10):
- Norway (10):
  - Medi3, Ålesund
  - Hodepineklinikkken Bergen, Bergen
  - Anub Mathew Thomas, Drammen
  - Helsa Fonna Trust, Haugesund
  - Møre og Romsdal Hospital Trust, Molde
  - Kristina Devik, Namsos
  - Oslo University Hospital, Oslo
  - Hodeverket, Sandnes
  - Sandvika Nevrosenter, Sandvika
  - St Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aamodt AH, Ueland T, Boldingh M, Bezgal BE, Argren MB, Dunne CA, Otterdal K, Gregersen I, Bjerkeli V, Michelsen AE, Husoy A, Morsund AH, Devik K, Poole AC, Gjendemsjo KB, Schluter K, Mathisen SM, Aalstad-Johansen M, Skattor TH, Sonnervik J, Boye TB, Popperud TH, Hogestol EA, Harbo HF, Lund-Johansen F, Aukrust P, Tronvik E, Dahl TB, Halvorsen BE. Altered amyloid plasma profile in patients with disabling headaches after SARS-CoV-2 infection and vaccination. BMJ Neurol Open. 2025 Aug 26;7(2):e001013. doi: 10.1136/bmjno-2024-001013. eCollection 2025. PMID 40881041